CLINICAL TRIAL: NCT01046669
Title: Evaluating the Use of Polymyxin B Hemoperfusion in a Randomized Controlled Trial of Adults Treated for Endotoxemia and Septic Shock
Brief Title: Safety and Efficacy of Polymyxin B Hemoperfusion (PMX) for Septic Shock
Acronym: EUPHRATES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spectral Diagnostics (US) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SDI-PMX-NA001
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Septic Shock; Endotoxemia
MeSH Terms: conditions — Shock, Septic; Endotoxemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Sham Comparator): Standard medical care for septic shock
  Interventions: Other: Standard medical care for septic shock
- Treatment (Experimental): Two (2) PMX cartridges will be administered approximately 24 hours apart plus standard medical care for septic shock
  Interventions: Device: TORAYMYXIN PMX-20R (PMX cartridge); Other: Standard medical care for septic shock

INTERVENTIONS:
Device: TORAYMYXIN PMX-20R (PMX cartridge) — TORAYMYXIN PMX-20R (PMX cartridge), Extracorporeal hemoperfusion device. Each treatment will target 2 hours with a minimum of 1 ½ hours, at a flow rate of approximately 100 ml/minute, (range of 80 to 120 ml/minute).
  Arms: Treatment
Other: Standard medical care for septic shock — Standard medical care for septic shock

SUMMARY:
To compare the safety and efficacy of the PMX cartridge based on mortality at 28-days in subjects with septic shock who have high levels of endotoxin and are treated with standard medical care plus use of the PMX cartridge, versus subjects who receive standard medical care alone.

ELIGIBILITY:
Inclusion Criteria:

* Hypotension requiring vasopressor support
* The subject must have received intravenous fluid resuscitation
* Documented or suspected infection
* Endotoxin Activity Assay ≥ 0.60 EAA units
* Evidence of at least 1 new onset organ dysfunction

Exclusion Criteria:

* Inability to achieve or maintain a minimum mean arterial pressure (MAP) of 65mmHg
* Subject has end stage renal disease and requires chronic dialysis
* There is clinical support for non-septic shock
* Subject has had chest compressions as part of CPR
* Subject has had an acute myocardial infarction (AMI)
* Subject has uncontrolled hemorrhage
* Major trauma within 36 hours of screening
* Subject has severe granulocytopenia
* HIV infection with a last known or suspected CD4 count of <50/mm3
* Subject has sustained extensive third-degree burns
* Body weight < 35 kg (77 pounds)
* Known hypersensitivity to polymyxin B
* Subject has known sensitivity or allergy to heparin
* Subject has screening MOD score of ≤9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Dellinger, Dr., Principal Investigator — Cooper Health System
Locations (40):
- United States (33):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Loma Linda, California
  - San Diego, California
  - Stanford, California
  - Colorado Springs, Colorado
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Augusta, Georgia
  - Idaho Falls, Idaho
  - Oak Park, Illinois
  - Peoria, Illinois
  - Iowa City, Iowa
  - Hazard, Kentucky
  - Baltimore, Maryland
  - Springfield, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Rochester, Minnesota
  - Jackson, Mississippi
  - St Louis, Missouri
  - Omaha, Nebraska
  - Camden, New Jersey
  - New York, New York
  - Greenville, North Carolina
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Chattanooga, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Richmond, Virginia
- Canada (7):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Victoria, British Columbia
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Québec, Quebec

REFERENCES:
- [Derived] Klein DJ, Foster D, Walker PM, Bagshaw SM, Mekonnen H, Antonelli M. Polymyxin B hemoperfusion in endotoxemic septic shock patients without extreme endotoxemia: a post hoc analysis of the EUPHRATES trial. Intensive Care Med. 2018 Dec;44(12):2205-2212. doi: 10.1007/s00134-018-5463-7. Epub 2018 Nov 23. PMID 30470853
- [Derived] Dellinger RP, Bagshaw SM, Antonelli M, Foster DM, Klein DJ, Marshall JC, Palevsky PM, Weisberg LS, Schorr CA, Trzeciak S, Walker PM; EUPHRATES Trial Investigators. Effect of Targeted Polymyxin B Hemoperfusion on 28-Day Mortality in Patients With Septic Shock and Elevated Endotoxin Level: The EUPHRATES Randomized Clinical Trial. JAMA. 2018 Oct 9;320(14):1455-1463. doi: 10.1001/jama.2018.14618. PMID 30304428
- [Derived] Klein DJ, Foster D, Schorr CA, Kazempour K, Walker PM, Dellinger RP. The EUPHRATES trial (Evaluating the Use of Polymyxin B Hemoperfusion in a Randomized controlled trial of Adults Treated for Endotoxemia and Septic shock): study protocol for a randomized controlled trial. Trials. 2014 Jun 11;15:218. doi: 10.1186/1745-6215-15-218. PMID 24916483

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 450 subjects randomized out of 921 clinically eligible subjects in 55 ICUs. First patient screened in Jun 2010, last patient screened in Jun 2016.
Pre-assignment Details: The following screened subjects were not randomized:
  * Subject's EAA <0.06 EA units
  * Subject met an exclusion criteria prior to randomization
  * Informed consent for the treatment phase of the study was not signed or consent withdrawn prior to randomization.
  Subjects who were randomized but not treated (RNT) were not part of safety analysis.
Groups:
- Sham: Standard medical care for septic shock
- Treatment: Two (2) PMX cartridges administered approximately 24 hours apart, plus standard medical care for septic shock.
Period: Overall Study
Arm/Group | Sham | Treatment
Started | 226 | 224
Completed | 226 | 223
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized subjects had baseline assessments completed
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham | Treatment | Total
Number analyzed (Participants) | 226 | 224 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (14.7) | 60.9 (15.1) | 59.8 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 84 | 177
  Male | 133 | 140 | 273
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 187 | 183 | 370
  Black | 13 | 22 | 35
  Hispanic | 12 | 10 | 22
  Asian | 9 | 3 | 12
  Other | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  Canada | 57 | 53 | 110
  United States | 169 | 171 | 340

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Compare mortality at 28 days in subjects treated with standard medical care plus PMX cartridge, versus subjects who received standard medical care alone
Time Frame: 28 days
Population: All subjects randomized
Measure: Count of Participants; unit: Participants
Groups:
- Treatment: Two (2) PMX cartridges administered approximately 24 hours apart plus standard medical care for septic shock
Arm/Group | Sham | Treatment
Number analyzed (Participants) | 226 | 224
Participants | 78 | 84

ADVERSE EVENTS:
Time Frame: Adverse events collected from Day 0 to Day 28. Serious adverse events (SAE, SADE, USADE) collected from Day 0 to 12 months post treatment.
Description: Subjects who were randomized but not treated (RNT) were not part of the safety analysis.
  12 out of 224 in the Treatment arm withdrew/were withdrawn prior to study treatment administration. Therefore, number of subjects at risk in this group is 212.
  6 out of 226 in the Sham arm withdrew/were withdrawn prior to sham procedure. Therefore, number of subjects at risk in this group is 220.
Arm/Group | Sham | Treatment
All-Cause Mortality (participants affected / at risk) | 78/226 | 84/224
Serious Adverse Events (participants affected / at risk) | 126/220 | 140/212
Other Adverse Events (participants affected / at risk) | 60/220 | 56/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham (N=220) | Treatment (N=212)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 6 (6) — 3 events on treatment arm possibly related to PMX cartridge
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (3)
Cardiac arrest (Cardiac disorders) | 12 (14) | 6 (6)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 8 (8) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 1 (2) | 0 (0)
Cor pulmonale chronic (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 3 (3) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Torsade de pointes (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal harmorrhage (Endocrine disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 5 (5)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstructive gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cardiac Death (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 6 (6)
Device leakage (General disorders) | 0 (0) | 1 (1) — 1 event on treatment arm probably related to PMX cartridge
Device malfunction (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 12 (12) | 14 (14)
Terminal state (General disorders) | 1 (1) | 0 (0)
Thrombosis in device (General disorders) | 0 (0) | 1 (1) — 1 event on treatment arm definitely related to PMX cartridge
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic hepatic failure (General disorders) | 2 (2) | 0 (0)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 4 (4)
Hepatic infarction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Biliary sepsis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 20 (23) | 23 (26)
Septic shock (Infections and infestations) | 16 (17) | 13 (13)
Splenic abscess (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Uninary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Wound sepsis (Infections and infestations) | 0 (0) | 1 (1)
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diaphragmatic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splenic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound evisceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood lactic acid increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adrenal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem stroke (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 2 (3)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Eating disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status change (Psychiatric disorders) | 1 (1) | 1 (1)
Faecaluria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 6 (6) | 3 (3)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Aspiration (Reproductive system and breast disorders) | 3 (4) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Epitaxis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 8 (10)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Purpura fulminans (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Steven-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (4)
Bleeding varicose vein (Vascular disorders) | 0 | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 2 (2)
Embolism (Vascular disorders) | 0 (0) | 2 (2)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (2) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 2 (2) — 2 events on treatment arm probably related to PMX cartridge
Infarction (Vascular disorders) | 1 (1) | 0 (0)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Vascular insufficiency (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham (N=220) | Treatment (N=212)
Cardiac arrest (Cardiac disorders) | 12 (14) | 6 (6)
Multi-organ failure (General disorders) | 12 (12) | 14 (14)
Sepsis (Infections and infestations) | 20 (23) | 23 (26)
Septic shock (Infections and infestations) | 16 (17) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor will be given a copy of the disclosure for review at least 60 days prior to the date of submission for publication or public disclosure. Sponsor may request to delete confidential information, other than study data. PI agrees to discuss with sponsor any of sponsor's suggestions with respect to the presentation of study data and the timing of the disclosure.